CLINICAL TRIAL: NCT03420170
Title: The Effects of Graded Exercise Integrated Education on Physical Fitness, Exercise Self-efficacy, and Physical Activity Level in People With Spinal Cord Injury
Brief Title: Physical Fitness, Exercise Self-efficacy, Physical Activity Level in People With Spinal Cord Injury (SCI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Noor Hafifi Noor Hisham, Principal Investigator, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universiti Teknologi MARA
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Spinal Cord Injuries; Physical Disability
Keywords: Spinal Cord Injuries; Physical Fitness; Exercise Self-Efficacy; Physical Activity
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Exercise Integrated Education (Experimental): The graded exercise (8 weeks)
  1. Strengthening exercise
  2. Aerobic Exercise
  Educational session to increase exercise self-efficacy and physical activity level (16 weeks)
  Interventions: Other: Graded Exercise Integrated Education
- Conventional physical therapy (Active Comparator): Normal routine of physical therapy (8 weeks)
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Graded Exercise Integrated Education — Aerobic exercise Wheelchair propelling, boxing, hand cycling (2 rounds)
  1. 3 mins. exercise and 2 mins. rest
  2. Increased to 4.5 mins. and 30 sec. rest
  Strengthening exercise:
  Vertical chest press, butterfly press; vertical row and wide lattissimus pull down 3 sets, 10 reps. and 2 min rest between sets, moderate to vigorous intensity (50% of 1 RM)
  Educational intervention:
  The educational intervention for exercise self-efficacy and physical activity level (2 hours a week for 8 weeks during in rehabilitation and once a month for 8 weeks after discharge from rehabilitation)
  Arms: Graded Exercise Integrated Education
Other: Conventional Physical Therapy — Normal routine of physical therapy including mobility training, wheelchair skills, resistance exercise, aerobic training, balance exercise, functional exercise
  Arms: Conventional physical therapy

SUMMARY:
This is a single blind randomized controlled trial study which will conducted on people with paraplegia wheelchair users. The objectives of this study is to investigates the effects of 16 weeks of 'Graded Exercise Integrated Education' over conventional physical therapy on physical fitness, exercise self-efficacy and the level of physical activity. There will be a significant difference between the experimental and control group.

DETAILED DESCRIPTION:
A study protocol will be a single blinded randomised controlled trial. 40 subjects with diagnosed of paraplegia (T1 and below) and dependent with wheelchair will be randomly assigned into 2 groups, Graded exercise (n=20) or Conventional Physical Therapy (n=20). In 8 weeks, the graded exercise group will receive strengthening and aerobic exercise for 2 times a week, and the controlled group will continue their normal routine. The strengthening exercise will consist of strength training for major upper limb muscles in the multigym station and free weights dumbbell whereas the aerobic exercise will perform by using arm ergometry, boxing and wheelchair wheeling. The exercise will be graded and progressed for each week in 8 weeks. The graded exercise group also will receive educational intervention to increase the exercise self-efficacy and physical activity level which will conduct in face to face for 2 times a week in 8 weeks during in-rehabilitation program and once on every 4 weeks in 8 weeks after discharge from in-rehabilitation program. The outcomes are the strength and endurance of upper limb which will be measure by using a BIODEX® Isokinetic Machine and hand grip strength by JAMAR® Hand-held dynamometry. The cardiovascular endurance will be measure by using 6 minute wheelchair push test (6MWPT). The exercise self-efficacy and physical activity level will be measure by using 'Exercise Self-Efficacy Scale (ESES)' and 'Physical Activity Scale for Individual with Disability (PASIPD)'. The outcome measure will be evaluated at the baseline level, week 4th, week 8th, week 12th, and 16th. Statistical analysis will be carried out using the SPSS 21.0 program for Windows and a significant level of p ≤ 0.05 will be used for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and Non-traumatic paraplegia
* Wheelchair dependent
* Age range between 18 and 65 years old

Exclusion Criteria:

* Pregnancy
* Individual who suffered from progressive neurological diseases, depression and mental disorder
* Individual with frequent autonomic dysreflexia and hypotension
* Individual with comorbid recent fracture
* Individual with severe heart diseases and pain
* Individual who not understand Malay and English
* Individual who not understand instructions and obey commands
* Individual who difficult to reach via telephone, email or social media

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular fitness | Change from baseline of cardiovascular endurance at 4 months
  6-Minute Wheelchair Push Test (6-MWPT)
Muscle strength | Change from baseline of upper limbs strength at 4 months
  The upper limb strength measure by using BIODEX ® Isokinetic machine
Muscle strength normalize with body weight | Change from baseline of upper limbs strength normalize body weight at 4 months
  The upper limb strength normalize with body weight measure by using BIODEX ® Isokinetic machine
Muscle endurance | Change from baseline of upper limbs endurance at 4 months
  The upper limb endurance measure by using BIODEX ® Isokinetic machine
Grip strength | Change from baseline of grip strength at 4 months
  The JAMAR ® hand held dynamometer
Exercise self-efficacy | Change from baseline of exercise self-efficacy at 4 months
  The Spinal Cord Injury Exercise Self-Efficacy (ESES)
Physical activity level | Change from baseline of physical activity level at 4 months
  The Physical Activity Scale for Individuals with Physical Disabilities (PASIPD)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hisham H, Justine M, Hussain H, Hasnan N, Manaf H. Effects of Graded Exercises Integrated with Education on Physical Fitness, Exercise SelfEfficacy, and Activity Levels in People with Spinal Cord Injury: A Quasi-Experimental Study Protocol. Asian Spine J. 2019 Mar 15;13(4):577-583. doi: 10.31616/asj.2018.0172. Print 2019 Aug. PMID 30866621